CLINICAL TRIAL: NCT04171466
Title: A Randomized, Double-blind, Placebo-controlled Study to Determine the Efficacy of a Multi-strain Synbiotic (SH-DS01) to Restore Gut Barrier Integrity and Gut Microbiota Composition After Antibiotic Administration.
Brief Title: Metagenomic and Metabolomic Reconstitution of Gut Microbiota After Broad Spectrum Antibiotic Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seed Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 19SAHS
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Antibiotic Side Effect; Antibiotic-associated Diarrhea; Antibiotic-induced Dysbiosis; Antibiotic-induced Epithelial Barrier Disintegrity
Keywords: Gut microbiome; Dysbiosis; Antibiotic therapy; Rationally-defined consortia; Short-chain fatty acids; Gut metabolome; Metagenomic sequencing; Ciproflozacin; Metronidazole; Probiotic Therapy
MeSH Terms: conditions — Dysbiosis | interventions — Ciprofloxacin; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Broad Spectrum Antibiotic Therapy + Microbial Consortia (Active Comparator)
  Interventions: Other: Ciprofloxacin + Metronidazole; Other: SH-DS01
- Broad Spectrum Antibiotic Therapy + Placebo (Placebo Comparator)
  Interventions: Other: Ciprofloxacin + Metronidazole; Other: Placebo
- No Antibiotic Therapy + Microbial Consortia (Active Comparator)
  Interventions: Other: SH-DS01
- No Antibiotic Therapy + Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Ciprofloxacin + Metronidazole — Participants will be instructed to take 1 capsule of Ciprofloxacin (500mg) twice daily for 7 days and 1 capsule of Metronidazole (500mg) thrice daily for 7 days. Antibiotics should be taken at least 2 hours before or 6 hours after mineral supplements containing magnesium or aluminum, as well as sucralfate, metal cations such as iron, and multivitamin preparations with zinc.
  Arms: Broad Spectrum Antibiotic Therapy + Microbial Consortia; Broad Spectrum Antibiotic Therapy + Placebo
Other: SH-DS01 — SH-DS01 is a rationally defined microbial consortia consisting of 24 strains across 12 species, with polyphenolic and phenolic prebiotic bioactive compounds. Participants will be instructed to take 2 capsules daily for the duration of the trial.
  Arms: Broad Spectrum Antibiotic Therapy + Microbial Consortia; No Antibiotic Therapy + Microbial Consortia
Other: Placebo — Placebo capsules for SH-DS01 will contain rice flour matched for color and texture in an identical outer capsule shell. Participants will be instructed to take 2 capsules daily for the duration of the trial.
  Arms: Broad Spectrum Antibiotic Therapy + Placebo; No Antibiotic Therapy + Placebo

SUMMARY:
In the United States, healthcare providers prescribe over 270 million antibiotic prescriptions each year. While antibiotics have transformed medicine and methods of treating life-threatening bacterial infection, broad spectrum antibiotics also induce disruption of resident gut microbial communities by altering both composition and function. This disruption of microbial community dynamics has been demonstrated at the taxonomic level, yet the extent of functional disruptions to microbial metabolic output and host cells remains understudied in humans. This study explores the impact of a broad spectrum antibiotic cocktail on microbial communities throughout the gastrointestinal tract, and the impact of a defined, multi-strain consortia of probiotic organisms following antibiotic exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Males & Females 18-55 years of age, inclusive
2. BMI of 18.5 - 29.9 kg/m2, inclusive
3. Waist circumference < 102 cm in males or < 88 cm in females
4. Female participant is not of child-bearing potential, defined as females who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, total endometrial ablation) Or, Females of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months.
5. Healthy as determined by laboratory results, medical history, and physical exam by QI
6. Agrees to abstain from use of fermented foods or beverages with live bacteria or products containing active cultures for the duration of the study
7. Agrees to avoid alcoholic beverages and drugs containing alcohol during antibiotic treatment period and for at least one day after (days 0-8)
8. Agrees to avoid high caffeine intake (no more than 1 cup of coffee or 300 mg of caffeine/day) during antibiotic treatment period of the study (days 0-7)
9. Agrees to refrain from intake of Nonsteroidal Anti-Inflammatory Drugs (NSAIDs) during antibiotic treatment period of the study (days 0-7) and 72 hours prior to prior to lactulose and mannitol test
10. Agrees to refrain from using drugs and supplements containing aluminum, magnesium, sorbitol and/or mannitol 72 hours prior to lactulose and mannitol test.
11. Agrees to comply with all study procedures
12. Agrees to maintain current level of physical activity throughout the study

Exclusion Criteria:

1. Women who are pregnant, breast feeding, or planning to become pregnant during the trial
2. Allergy or sensitivity to antibiotics (Ciprofloxacin, Metronidazole), Lactulose or Mannitol, or investigational product's active or inactive ingredients
3. Use of antibiotics or antifungals within three months prior to enrollment, including topical antibiotics or antifungals.
4. Clinically significant abnormal laboratory results at screening as assessed by the QI
5. Use of PPIs and H2-antagonists
6. Use of tobacco products
7. Type I or type II diabetes mellitus or treatment with anti-diabetic medication
8. Unstable metabolic diseases or chronic diseases as assessed by the QI
9. Self-reported current or pre-existing thyroid condition.
10. Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
11. Current or history of any significant diseases of the gastrointestinal tract that may impact study outcomes as assessed by the QI
12. Significant cardiovascular event in the past 6 months. If the event occurred greater that 6 months ago and if on stable medication may be included after assessment by the QI on a case by case basis
13. Major surgery in the past 3 months or individuals who have planned surgery during the course of the trial. Participants with minor surgery will be considered on a case-by-case basis by the QI
14. Self-reported an autoimmune disease or an immune-compromised state
15. Self-reported HIV-, Hepatitis B- and/or C-positive diagnosis
16. History of or current diagnosis with kidney and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones symptom free for 6 months
17. Self-reported medical or neuropsychological condition and/or cognitive impairment that, in the QI's opinion, could interfere with study participation
18. Self-reported blood/bleeding disorder. To be confirmed by the QI on a case by case basis
19. Cancer in the five years prior to enrollment, except skin cancers completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable following case by case assessment by QI.
20. Clinically significant illness in the four weeks prior to randomization
21. Current use of prescribed medications listed in Section 7.3.1
22. Current use of over-the-counter medications, supplements, foods and/or drinks listed in Section 7.3.2
23. Current use of any probiotic, prebiotic and symbiotic product unless willing to undergo a 4-week washout and abstain from consuming such products during the study.
24. Medical use of cannabinoid products
25. Use of any cannabinoid products (including synthetics) within one month of study entry
26. Alcohol or drug abuse within the last 12 months
27. High alcohol intake (>2 per day or a total of >10 standard drinks per week)
28. Blood donation 30 days prior to screening, during the study, or a planned donation within 30-days of the last study visit
29. Participation in other clinical research trials 30 days prior to screening
30. Any other active or unstable medical condition, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Change in microbiota composition at 3 months as assessed by whole genome shotgun sequencing. | Baseline- Days 91
  Microbiota composition will be identified through fecal samples for total genomic DNA extraction in participants supplemented with SH-DS01 and with or without antibiotics.

SECONDARY OUTCOMES:
Difference in serum LPS-binding protein (LBP) at Day 7. | Baseline- Days 91
  As a measure of intestinal barrier integrity in response to antibiotic therapy.
Difference in the Intestinal Permeability Assessment (IPA) at Day 7 as measured by Lactulose/mannitol testing. | Baseline- Days 91
  As a measure of intestinal barrier integrity in response to antibiotic therapy.
Metabolomic profile of stool samples. | Baseline- Days 91
  As assessed by untargeted metabolomics on whole stool samples.
Number of participants with improved Antibiotic-Associated Gastrointestinal Function | Baseline- Days 91
  As assessed by daily symptom tracking software of stool quality, regularity, ease of expulsion, bloating, flatulence, and intestinal transit time.

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Reid, PhD, Principal Investigator — Lawson Health Research Institute, St. Joseph's Hospital
Locations (1):
- KGK Science, London, Ontario, Canada

REFERENCES:
- [Background] Qin J, Li R, Raes J, Arumugam M, Burgdorf KS, Manichanh C, Nielsen T, Pons N, Levenez F, Yamada T, Mende DR, Li J, Xu J, Li S, Li D, Cao J, Wang B, Liang H, Zheng H, Xie Y, Tap J, Lepage P, Bertalan M, Batto JM, Hansen T, Le Paslier D, Linneberg A, Nielsen HB, Pelletier E, Renault P, Sicheritz-Ponten T, Turner K, Zhu H, Yu C, Li S, Jian M, Zhou Y, Li Y, Zhang X, Li S, Qin N, Yang H, Wang J, Brunak S, Dore J, Guarner F, Kristiansen K, Pedersen O, Parkhill J, Weissenbach J; MetaHIT Consortium; Bork P, Ehrlich SD, Wang J. A human gut microbial gene catalogue established by metagenomic sequencing. Nature. 2010 Mar 4;464(7285):59-65. doi: 10.1038/nature08821. PMID 20203603
- [Background] Korpela K, Salonen A, Vepsalainen O, Suomalainen M, Kolmeder C, Varjosalo M, Miettinen S, Kukkonen K, Savilahti E, Kuitunen M, de Vos WM. Probiotic supplementation restores normal microbiota composition and function in antibiotic-treated and in caesarean-born infants. Microbiome. 2018 Oct 16;6(1):182. doi: 10.1186/s40168-018-0567-4. PMID 30326954
- [Background] De Wolfe TJ, Eggers S, Barker AK, Kates AE, Dill-McFarland KA, Suen G, Safdar N. Oral probiotic combination of Lactobacillus and Bifidobacterium alters the gastrointestinal microbiota during antibiotic treatment for Clostridium difficile infection. PLoS One. 2018 Sep 28;13(9):e0204253. doi: 10.1371/journal.pone.0204253. eCollection 2018. PMID 30265691
- [Background] Kristensen NB, Bryrup T, Allin KH, Nielsen T, Hansen TH, Pedersen O. Alterations in fecal microbiota composition by probiotic supplementation in healthy adults: a systematic review of randomized controlled trials. Genome Med. 2016 May 10;8(1):52. doi: 10.1186/s13073-016-0300-5. PMID 27159972
- [Background] Rodgers B, Kirley K, Mounsey A. PURLs: prescribing an antibiotic? Pair it with probiotics. J Fam Pract. 2013 Mar;62(3):148-50. PMID 23520586
- [Background] Nagpal R, Wang S, Ahmadi S, Hayes J, Gagliano J, Subashchandrabose S, Kitzman DW, Becton T, Read R, Yadav H. Human-origin probiotic cocktail increases short-chain fatty acid production via modulation of mice and human gut microbiome. Sci Rep. 2018 Aug 23;8(1):12649. doi: 10.1038/s41598-018-30114-4. PMID 30139941
- [Background] Smith PM, Howitt MR, Panikov N, Michaud M, Gallini CA, Bohlooly-Y M, Glickman JN, Garrett WS. The microbial metabolites, short-chain fatty acids, regulate colonic Treg cell homeostasis. Science. 2013 Aug 2;341(6145):569-73. doi: 10.1126/science.1241165. Epub 2013 Jul 4. PMID 23828891
- [Background] Cox MA, Jackson J, Stanton M, Rojas-Triana A, Bober L, Laverty M, Yang X, Zhu F, Liu J, Wang S, Monsma F, Vassileva G, Maguire M, Gustafson E, Bayne M, Chou CC, Lundell D, Jenh CH. Short-chain fatty acids act as antiinflammatory mediators by regulating prostaglandin E(2) and cytokines. World J Gastroenterol. 2009 Nov 28;15(44):5549-57. doi: 10.3748/wjg.15.5549. PMID 19938193
- [Background] Ho L, Ono K, Tsuji M, Mazzola P, Singh R, Pasinetti GM. Protective roles of intestinal microbiota derived short chain fatty acids in Alzheimer's disease-type beta-amyloid neuropathological mechanisms. Expert Rev Neurother. 2018 Jan;18(1):83-90. doi: 10.1080/14737175.2018.1400909. Epub 2017 Nov 14. PMID 29095058
- [Background] Resta-Lenert S, Barrett KE. Probiotics and commensals reverse TNF-alpha- and IFN-gamma-induced dysfunction in human intestinal epithelial cells. Gastroenterology. 2006 Mar;130(3):731-46. doi: 10.1053/j.gastro.2005.12.015. PMID 16530515
- [Background] van Baarlen P, Troost F, van der Meer C, Hooiveld G, Boekschoten M, Brummer RJ, Kleerebezem M. Human mucosal in vivo transcriptome responses to three lactobacilli indicate how probiotics may modulate human cellular pathways. Proc Natl Acad Sci U S A. 2011 Mar 15;108 Suppl 1(Suppl 1):4562-9. doi: 10.1073/pnas.1000079107. Epub 2010 Sep 7. PMID 20823239
- [Background] Suez J, Zmora N, Zilberman-Schapira G, Mor U, Dori-Bachash M, Bashiardes S, Zur M, Regev-Lehavi D, Ben-Zeev Brik R, Federici S, Horn M, Cohen Y, Moor AE, Zeevi D, Korem T, Kotler E, Harmelin A, Itzkovitz S, Maharshak N, Shibolet O, Pevsner-Fischer M, Shapiro H, Sharon I, Halpern Z, Segal E, Elinav E. Post-Antibiotic Gut Mucosal Microbiome Reconstitution Is Impaired by Probiotics and Improved by Autologous FMT. Cell. 2018 Sep 6;174(6):1406-1423.e16. doi: 10.1016/j.cell.2018.08.047. PMID 30193113
- [Background] Spiller RC. Hidden Dangers of Antibiotic Use: Increased Gut Permeability Mediated by Increased Pancreatic Proteases Reaching the Colon. Cell Mol Gastroenterol Hepatol. 2018 Jul 11;6(3):347-348.e1. doi: 10.1016/j.jcmgh.2018.06.005. eCollection 2018. No abstract available. PMID 30182044